CLINICAL TRIAL: NCT05760092
Title: The Use of Photobiomodulation in the Treatment of Oral Complaints of Long COVID-19. A Randomized Controlled Trial.
Brief Title: The Use of Photobiomodulation in the Treatment of Oral Complaints of Long COVID-19.A Randomized Controlled Trial.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Rebeca Boltes Cecatto, Professor at Post-Graduate Program of Biophotonics Applied at Health Sciences, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Covidlongasusy
Record Dates: First submitted 2022-09-20; First posted 2023-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Xerostomia; COVID-19; Long COVID; Persistent COVID-19
Keywords: Xerostomia; Dry Mouth; COVID-19; Long Covid; Photobiomodulation
MeSH Terms: conditions — Xerostomia; COVID-19; Post-Acute COVID-19 Syndrome | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation Therapy (Experimental): Institutional standard treatment for xerostomia and COVID Longa + PBM therapy
  Interventions: Combination Product: Institutional standard treatment for xerostomia and Long Covid; Radiation: Photobiomodulation Therapy
- Placebo Photobiomodulation (Placebo Comparator): Institutional standard treatment for xerostomia and COVID Longa + PBM placebo therapy
  Interventions: Combination Product: Institutional standard treatment for xerostomia and Long Covid; Radiation: Placebo Photobiomodulation Therapy

INTERVENTIONS:
Combination Product: Institutional standard treatment for xerostomia and Long Covid — (Medical follow-up at the general outpatient clinic for prescription and control of medications, underlying diseases, clinical status and routine short, medium and long-term care follow-up, standard guidelines for the use of aerobic physical activity in those who do not have contraindications, stretching exercises, ergonomics, home adaptation to maximize functionality and energy savings, emotional cognitive support psychotherapy, socio-educational measures, sleep hygiene, Nutritional follow-up and monitoring, dentistry follow-up at the University's odontological team, guidance on proper oral hygiene, use of low-sugar diets, daily topical use of fluoride and antimicrobial mouthwash to prevent dental caries, oral hydration, guidance on avoiding cigarette use or intake of caffeine-containing beverages . When necessary, measures such as oral lubricants, artificial saliva, measures to prevent aspirations, as well as the careful use of liquids during meals, can be instituted ) +
Radiation: Photobiomodulation Therapy — Application of Red LED in the 3 pairs of major salivary glands (parotid, submandibular and sublingual) extraorally, transcutaneously, for 36 seconds, twice a week for 06 weeks.
  Other Names: PBM therapy
  Arms: Photobiomodulation Therapy
Radiation: Placebo Photobiomodulation Therapy — All parameters as the number of points, dose and place of application of the PBM will be the same as described in the item PBM therapy Intervention Group, however in the placebo PBM equipment will be turned off. The device activation noise will be recorded and used to mimic the irradiation.
  Arms: Placebo Photobiomodulation

SUMMARY:
Coronavirus (COVID-19) is a newly emerging zoonotic agent that emerged in December 2019 in China (2019-nCoV) as a Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV -2). Long COVID-19, or Post-Covid Syndrome or Long-term COVID-19, is a post-viral syndrome that persists after the acute infection has resolved. The most frequent symptoms of Lonf-term COVID are fatigue and dyspnea. But two classes of symptoms have been received scientific attention: the musculoskeletal pain and oral complaints related to Long COVID, mainly xerostomia and burning mouth. Photobiomodulation (PBM) therapy is often used for oral diseases and presents itself as a non-invasive, low-cost, safe therapy that has benefits in relation to the quality of life of patients with xerostomia. This study aims to investigate the clinical effectiveness of the use of a Photobiomodulation protocol in the treatment xerostomia and oral complaints related to Long-Covid. This will be a single-center, randomized, controlled, blinded clinical trial that will involve patients with Long COVID in follow-up at the Medical and Multiprofessional outpatient clinic of University Nove de Julho (UNINOVE) which remained hospitalized with COVID-19 at Lydia Storópoli Universitarian Hospital during the year 2022 and who were discharged from the inpatient treatment from January to December 2022. All those patients presenting xerostomia, burning mouth or oral complaints related to Long Covid will be randomized into 2 groups: PBM Group (standard rehabilitation treatment for Long COVID and xerostomia + PBM therapy) or PBM placebo group (standard rehabilitation treatment for Long COVID and xerostomia + placebo PBM therapy). PBM consists of the application of Red LED on the 3 pairs of major salivary glands (parotid, submandibular and sublingual) extraorally, transcutaneously, 3 J/cm2, for 36 seconds, twice a week for 06 weeks. Functional and quality of life evaluations will be perform pre and post therapy period.

DETAILED DESCRIPTION:
Coronavirus (COVID-19) is a newly emerging zoonotic agent that emerged in December 2019 in China (2019-nCoV) and which results in Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV -2) The scientific literature has made progress in the characterization of the new coronavirus and works extensively on therapies and vaccines against the virus. However, it is now known that SARS-CoV-2 is more than just an acute respiratory syndrome. Long-term COVID-19, or Post-Covid Syndrome or Long-term COVID-19, is a post-viral syndrome that was first reported online in groups of COVID-19 survivors discussing their symptoms after the acute infection has resolved. It begins to gain recognition in the scientific and medical communities. Although a universally accepted definition does not yet exist, reviews have identified that the most frequent symptoms of Lonf-term COVID are fatigue and dyspnea. But two classes of symptoms have been received scientific attention: the musculoskeletal pain and xerostomia. Xerostomia is defined as a subjective sensation of dry mouth described by patients and which is commonly related to hyposalivation (decreased salivary flow rate). The pathophysiology and clinical evolution of xerostomia in COVID-19 still lacks studies, but there are reports of 2 to 30% of patients presenting the complaint of dry mouth sensation even after the resolution of acute COVID. Regular physical therapy, cognitive behavioral therapy have been used and encouraged in the follow-up of patients with post- COVID, demonstrating that even today these practices seem to be more promising than pharmacological treatment. In parallel, studies demonstrate that Photobiomodulation (PBM) therapy is often used for oral diseases and presents itself as a non-invasive, low-cost, safe therapy that has benefits in relation to the quality of life of these patients. PBM refers to a series of therapies in which non-ionizing light beams, including lasers, LEDs and broadband light in the visible and infrared spectra, are used to interact with biological tissues for different purposes. In this sense, this study aims to investigate the clinical effectiveness of the use of a Photobiomodulation protocol in the treatment xerostomia related to Long-Covid. This will be a single-center, randomized, controlled, blind clinical trial that will involve patients with Long-COVID in follow-up at the Medical and Multiprofessional outpatient clinic of University Nove de Julho (UNINOVE). An analysis will be carried out of all medical records of patients who remained hospitalized with COVID-19 at Lydia Storópoli Universitary Hospital during the year 2022 and who were discharged from the inpatient treatment from January to December 2022, for a survey of telephone contact and epidemiological data collection by medical records. All those patients who answer the questions referring to one or more symptoms related to the oral or nasal cavity, which have arisen after the onset of acute COVID infection, will be invited to participate in the study by making a first face-to-face evaluation at the University to confirm the diagnostic criteria of xerostomia, the diagnosis of Long COVID and evaluation of inclusion criteria in the study (adults with COVID-19 with complaints of xerostomia diagnosed more than 4 weeks after the acute infection and persisting for at least 02 months). Pre- and post-treatment evaluations are composed by the Brazilian Version of the SF 36 Quality of Life Scale, salivary sialometry and salivary pH, Oral Health Impact Profile (OHIP-14), Abbreviated Xerostomia Inventory (SXI), Brazilian version of the Functional Independence Measure (FIM), Post -Covid-19 Functional Status Scale and WHO Disability Assessment Scale (WHODAS 2.0) All patients included will be randomized into 2 groups: PBM Group (standard rehabilitation treatment for Long COVID and xerostomia + PBM therapy) or PBM placebo group (standard rehabilitation treatment for Long COVID and xerostomia + placebo PBM therapy). PBM consists of the application of Red LED on the 3 pairs of major salivary glands (parotid, submandibular and sublingual) extraorally, transcutaneously, 3 J/cm2, for 36 seconds, twice a week for 06 weeks. The results will be sent for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis xerostomia related to Long-COVID;
* more than 4 weeks after the acute infection hat have persisted for at least 02 months (regardless of whether these patients are already using treatment for the complaints or not);
* Age greater than 18 years.

Exclusion Criteria:

* Clinical diagnosis of other previous rheumatological or musculoskeletal diseases that presents xerostomia;
* Previous use in the last 90 days of laser treatment or other photobiomodulation technique for the same or another indication;
* Clinical manifestations or complaints of xerostomia related to diseases other than Long COVID;
* Previous diseases of the oral or nasal cavity that occur with the symptom of xerostomia;
* Systemic inflammatory diseases (rheumatoid arthritis, Reiter's arthritis, ankylosing spondylitis, generalized polyarthritis, neoplasms);
* Uncontrolled metabolic or endocrine diseases;
* Neoplastic diseases;
* Serious cognitive or psychiatric disorders that that do not allow the understanding of the study;
* Steroid injections during the last 48 hours prior to baseline study assessment;
* Use of corticosteroids at an immunosuppressive dose (20mg daily of prednisone or equivalent for at least 14 days);
* Infection or tumor at the site of therapy application;
* Current chronic infections such as tuberculosis or chronic hepatitis treated or not;
* Severe blood dyscrasia;
* Blood clotting disorders (including thrombosis) at the application site;
* Psychoaffective disorder that prevents adherence to treatment;
* Signs, symptoms or laboratory changes suggestive of acute reinfection by COVID 19;
* Elevated resting heart rate (>100 beats/min);
* Low or high blood pressure (<90/60 or >140/90 mmHg);
* Low blood oxygen saturation (<95%) at rest, or dyspnea grade 3, 4, or 5 on the Medical Research Council Dyspnea Scale (KOVELIS et al., 2008), or exacerbation of dyspnea on exertion;
* Any condition where exercise is a contraindication such as decompensated heart disease, decompensated diabetes;
* Contraindications to the rehabilitation treatment of post-COVID syndrome recommended by the WHO: presence of heart disease after acute COVID, decrease in blood oxygen saturation after exercise (below 94% or decrease of at least 3% of the baseline saturation), presence of orthostatic hypotension;
* Any photosensitive disease or light sensitivity condition;
* Loss of follow-up at the follow-up clinical outpatient clinic, despite maintaining use of PBM according to the study protocol;
* Pregnancy;
* Any adverse effect on the previous use of PBM.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Brazilian version of the SF 36 Quality of Life Scale | pre-treatment and post-treatment moment (after 04 weeks of treatment)
  Assessment of general quality of life, translated and validated for the Brazilian population, composed of assessments in the following domains: functional capacity, limitation due to physical aspects, pain, general health status, vitality, social aspects, emotional aspects and mental health.
Nutritional assessment | pre-treatment and post-treatment (after 04 weeks of treatment)
  Anthropometric measurements of body weight, height and calculation of the Body Mass Index (BMI) according to the World Health Organization (WHO) reference standard for adults and Lipschitz criterion for elderly patients.
Salivary ph, Stimulated salivary flow and unstimulated salivary flow | pre-treatment and post-treatment (after 04 weeks of treatment)
  Total salivary flow rates (SFRs) at rest and during stimulation will be determined according to the guidelines for unstimulated and stimulated total saliva collection provided by Navazesh and Kumar (1993). To characterize hyposalivation, investigators will use the Sreebny criterion (2000) according to which the abnormal salivary flow is lower than 0.1 ml/min without stimulation and 0.5 ml/min with stimulation. Salivary pH (unstimulated salivary flow) will also be evaluated, which will be performed using pH indicator paper tape, color scale ranging from 0.0 to 14.0 (gradation 1.0; precision 0.2) The strips will be dipped in samples of saliva for 5 min. Then the test fields of the strips will be compared with the color scales. Whereas healthy saliva must have a pH between 6.5 to 7.4.
Oral Health Impact Profile (OHIP-14) | pre-treatment and post-treatment (after 04 weeks of treatment)
  Assessment of Oral Health-related Quality of Life, by OHIP-14 , translated and validated for Brazilian population
Xerostomia Inventory XI | pre-treatment and post-treatment (after 04 weeks of treatment)
  A multi-item approach to measuring and quantify dry mouth.
Functional Independence Measure (FIM) | pre-treatment and post-treatment (after 04 weeks of treatment)
  A translated and validated for the Brazilian population of general assessment of functional independence
Post-Covid-19 Functional Status Scale | pre-treatment and post-treatment (after 04 weeks of treatment)
  A tool to measure the full spectrum of functional outcomes following COVID-19.
The World Health Organization Disability Assessment Schedule (WHODAS 2.0) | pre-treatment and post-treatment (after 04 weeks of treatment)
  The World Health Organization Disability Assessment Schedule (WHODAS 2.0) was designed to assess the functioning level in six life domains (cognition, mobility, selfcare, getting along, life activities, and participation in community activities)

CONTACTS AND LOCATIONS:
Overall Officials: Rebeca B Cecatto, M.D., Ph.D., Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho / Post-Graduate program Biophotonics Applied to Health Sciences, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chowdhury F, Grigoriadou S, Bombardieri M. Severity of COVID-19 infection in primary Sjogren's syndrome and the emerging evidence of COVID-19-induced xerostomia. Clin Exp Rheumatol. 2021 Nov-Dec;39 Suppl 133(6):215-222. doi: 10.55563/clinexprheumatol/k7x3ta. Epub 2021 Dec 16. PMID 34919045
- [Result] Verma H, Shah J, Akhilesh K, Shukla B. Patients' perspective about speech, swallowing and hearing status post-SARS-CoV-2 (COVID-19) recovery: E-survey. Eur Arch Otorhinolaryngol. 2022 May;279(5):2523-2532. doi: 10.1007/s00405-021-07217-2. Epub 2022 Jan 21. PMID 35059791